CLINICAL TRIAL: NCT06161935
Title: A Retrospective Study of Lymph Node Metastatic Pattern Based Incorporating Tumor Location, GGO Components and Size for Non-small Cell Lung Cancer Involving Patients in Thoracic Surgery Fudan University Shanghai Cancer Center From April 2008 to July 2022. Data Were Analyzed From October 2022 to July 2023 to Further Elaborated the Different Nodal Metastatic Pattern in Different Tumors and Identify the Characteristics of Patient Group Without Lymph Node Metastasis.
Brief Title: A Study of Lymph Node Metastatic Pattern Based Incorporating Tumor Location, GGO Components and Size for Non-small Cell Lung Cancer
Status: Completed | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Penghao Deng, Principal Investigator, Fudan University
Other Study IDs: JCY001
Record Dates: First submitted 2023-11-22; First posted 2023-12-08 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Lung Cancer Non Small Cell
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — no intervention, it is a retrospective study .

SUMMARY:
The goal of this observational study is to learn about in invasive non-small cell lung cancer patients who underwent pulmonary resection with systematic lymph node dissection from April 2008 to July 2022 . The main question it aims to answer are: determine the situation of zero risk mediastinal lymph metastases and the different lymph node metastatic patterns of tumors with different characteristics.

Participants will provide personal information to analyze. and there is not a comparison group.

ELIGIBILITY:
Inclusion Criteria:

* invasive non-small cell lung cancer patients in FUSCC who underwent pulmonary resection with systematic lymph node dissection from April 2008 to July 2022

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 7067 invasive non-small cell lung cancer patients in FUSCC who underwent pulmonary resection with systematic lymph node dissection from April 2008 to July 2022.
Sampling Method: Non-Probability Sample
Enrollment: 7067 (Actual)
Dates: Start 2008-04 (Actual); Primary Completion 2022-07 (Actual); Study Completion 2023-07 (Actual)

PRIMARY OUTCOMES:
The number of participants with no mediastinal lymph metastases after systematic lymph node dissection. | 1 year
  We counted the number of participants with no mediastinal lymph metastases after systematic lymph node dissection and tried to determine the situation of zero risk mediastinal lymph metastases after our analyses.